CLINICAL TRIAL: NCT04670172
Title: Real-Life Chronic Rhinosinusitis Outcome Registry
Status: Recruiting | Type: Observational
Sponsor: Change Accelerator in Respiratory Care (Industry)
Responsible Party: Sponsor
Other Study IDs: GHOR001
Record Dates: First submitted 2020-11-25; First posted 2020-12-17 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic rhinosinusitis patients: Adult chronic rhinosinusitis patients capable of using a mobile application.

SUMMARY:
An international consortium of leading medical experts in the field of chronic respiratory disease, the research team of Galenus Health and the non-profit organization EUFOREA (European Forum for Research and Education in Allergy and Airway diseases) has been conceived to conduct real-life outcome research. The Galenus Health digital platform consisting of a mobile application for patients and an online dashboard for physicians will be implemented in each of the participating centres. The data will be centralized in a pseudonymized database and will be the basis of the Chronic RhinoSinusitis Outcome Registry.

DETAILED DESCRIPTION:
This real-life chronic rhinosinusitis outcome registry aims at longitudinal data collection from patients attending specialist care centres across Europe.

As primary aim it intends to provide new insights on the burden of uncontrolled disease, the impact on health-related quality of life, productivity loss as well as the effect of disease severity and co-morbid disease on these outcome parameters.

In addition this outcome registry intends to identify patients eligible for type 2 targeted biologic therapy, evaluate treatment effectiveness and markers of treatment response.

Beyond that direct and indirect costs for society related to chronic rhinosinusitis and its' treatment will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of Chronic RhinoSinusitis
* Capable of using a mobile application on a smartphone

Exclusion Criteria:

* Patients with malignancies of the sinonasal cavity
* Patients with inverted papilloma
* Patients with unilateral disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Users of the Galenus Health mobile application who reported a diagnosis with CRS will be entered into the registry if they provided consent for scientific research. Confirmation of CRS diagnosis by a physician will be performed via the web-based dashboard. The CRS population includes both patients with and without nasal polyps, with and without asthma co-morbidity, with or without former surgery, aged 18 years or above. Patients are included into the registry with the aim of longitudinal follow up.
Sampling Method: Probability Sample
Enrollment: 4550 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom severity total symptoms | 1 year
  Baseline and change in VAS (visual analogue scale) total nasal, sinus, lung symptoms; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm

SECONDARY OUTCOMES:
Symptom severity - facial pain | 1 year
  Baseline and change in VAS facial pain; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - impaired smell | 1 year
  Baseline and change in VAS impaired smell; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - nasal blockage | 1 year
  Baseline and change in VAS nasal blockage; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - nasal secretions | 1 year
  Baseline and change in VAS nasal secretions; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - post-nasal drip | 1 year
  Baseline and change in VAS post-nasal drip; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - wheeze | 1 year
  Baseline and change in VAS post-nasal drip; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - dyspnoea | 1 year
  Baseline and change in VAS dyspnoea; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - chest tightness | 1 year
  Baseline and change in VAS chest tightness; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - cough | 1 year
  Baseline and change in VAS cough; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - itchy nose | 1 year
  Baseline and change in VAS itchy nose; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - itchy eyes | 1 year
  Baseline and change in VAS itchy eyes; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Symptom severity - sneeze | 1 year
  Baseline and change in VAS sneeze; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Disease impact - work or school | 1 year
  Baseline and change in VAS work or school; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Disease impact - sleep quality | 1 year
  Baseline and change in VAS impact sleep quality; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Disease impact - daily life activities | 1 year
  Baseline and change in VAS impact daily life activities; 0 (Not at all bothersome) - 100 (Extremely bothersome) mm
Healthcare utilisation | Registration at time of event
  Number of care pathway events (healthcare provider visits, emergency room visits, hospitalisation, CT scan, endoscopic sinus surgery, bronchial thermoplastic, diagnostic tests)
Medication use | Registration at time of new prescription and intakes
  Changes in medication
General health-related quality of life | 1 year
  EQ-5D-5L (EuroQol-5Dimension-5Level) questionnaire
CRS-specific quality of life | 1 year
  SNOT-22 (SinoNasal Outcome Test-22) questionnaire
Nasal Polyp Score | 1 year
  Baseline and change in nasal polyp score
Lund-Mackay score | 1 year
  Baseline Lund-Mackay score
Blood eosinophil counts | 1 year
  cells/mm^3
Serum total IgE | 1 year
  IU/ml
Work Performance and Activity Impairment | 1 year
  Work Performance and Activity Impairment questionnaire
Hospitalisations | 1 year
  Number of hospitalisation for nose, sinus or lung problem in the past year
Oral corticosteroid use | 1 year
  Courses of oral corticosteroid in the past year

CONTACTS AND LOCATIONS:
Overall Officials: Sven F Seys, PhD, Study Director — Change Accelerator in Respiratory Care; Claus Bachert, MD, PhD, Principal Investigator — UZ Ghent
Locations (13):
- Austria (2):
  - Graz University Hospital, Graz
  - University Hospital Vienna, Vienna
- Belgium (3):
  - UCL Saint-Luc, Brussels
  - UZ Ghent, Ghent
  - UZ Leuven, Leuven
- Odense University Hospital, Odense, Denmark
- Helsinki University Hospital, Helsinki, Finland
- CHU Lille, Lille, France
- Dusseldorf University Clinic, Düsseldorf, Germany
- Policlinico Umberto I, Rome, Italy
- UMC Amsterdam, Amsterdam, Netherlands
- Hospital Clinic de Barcelona, Barcelona, Spain
- Prof Claire Hopkins private practice, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided